CLINICAL TRIAL: NCT02086656
Title: PERIOPERATIVE TREATMENT WITH COI-B (CAPECITABINE, OXALIPLATIN, IRINOTECAN AND BEVACIZUMAB) OF HIGH RISK OR BORDERLINE RESECTABLE COLORECTAL CANCER LIVER METASTASES
Acronym: COI-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Filippo Pietrantonio, M.D., MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COI-B
Record Dates: First submitted 2013-12-20; First posted 2014-03-13 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer Liver Metastases
Keywords: liver metastases; colorectal cancer; perioperative treatment
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Experimental): Single arm, open label
  Interventions: Drug: capecitabine, oxaliplatin, irinotecan and bevacizumab

INTERVENTIONS:
Drug: capecitabine, oxaliplatin, irinotecan and bevacizumab — perioperative COI-B

SUMMARY:
Capecitabine, oxaliplatin, irinotecan and bevacizumab as perioperative strategy of borderline and/or high risk resectable colorectal cancer liver metastases

DETAILED DESCRIPTION:
Previous studies demonstrated a significant association between tumor regression grade of hepatic colorectal metastases (TRG1: complete pathological response; TRG2: major pathological response; TRG3: partial pathological response; versus TRG4-5 no pathological response) and outcome in terms of survival after neoadjuvant treatment. In particular, retrospective data showed an association between oxaliplatin-based chemotherapy and improvement of grade and percentage of tumor regression; moreover, the addition of Bevacizumab seems to improve TRG over chemotherapy alone, conferring also a protection against liver damage due to chemotherapy-induced sinusoidal obstruction syndrome.

This is the rationale that induced us to carry out an evaluation and feasibility assessment of a perioperative approach with COI-B regimen in patients affected by high risk or borderline resectable colorectal liver metastases, with or without previous resection of primary tumor.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Histological diagnosis of colorectal adenocarcinoma.
* Liver-limited metastases or metastases mainly (≥80% total disease burden) limited to the liver with extrahepatic disease judged resectable concomitantly or sequentially. Primary tumor may be resected or not, but patient must not be symptomatic for T.
* Previous adjuvant therapy is allowed if it had been terminated for at least 6 months.
* Previous first line treatment (irinotecan or oxaliplatin containing regimen) with stable or partial response after no more than 3 months of treatment
* Age >= 18 years
* Performance Status (ECOG <2)
* Adequate organ function including the following:
* Adequate bone marrow reserve: WBC count >3.0x109/L, absolute neutrophil count >1.5x109/L, platelet count >100x109/L, and hemoglobin >10 g/dL .
* Hepatic: bilirubin < 1.5 times the ULN, alkaline phosphatase, aspartate transaminase, and alanine transaminase < 2.5 xULN
* Renal : serum creatinin <2.0xULN
* Patients compliance and geographic proximity that allows for adequate follow-up
* Patients must sign an informed consent document (ICD)
* Male and female patients with reproductive potential must use an approved contraceptive method.

Exclusion Criteria:

* Tumor involvement of liver > 75%
* Chance of a liver remnant after surgery < 25%
* Eligibility for concurrent radiotherapeutic treatment
* Disease progression during first line chemotherapy with FOLFOX, XELOX, FOLFIRI or XELIRI plus bevacizumab
* Previous treatment with more than 3 months of FOLFOX or FOLFIRI
* Previous therapy with bevacizumab or cetuximab or panitumumab
* Administration of other experimental drugs during the study.
* Body Mass Index > 35
* Brain metastases.
* Pregnancy and breast-feeding.
* Serious or uncontrolled medical pathologies or active infections that would jeopardize the possibility of receiving the investigated treatment. Disorders that could influence the absorption of capecitabine (e.g. malabsorption), intestinal occlusion, Crohn's disease or ulcerative colitis.
* Psychiatric disorders, neurologic disease or other conditions that would make it impossible to comply with the protocol procedures. Peripheral neuropathy not related to oxaliplatin previous administration.
* Previous dangerous life threatening toxicities from fluoropyrimidine.
* Positive anamnesis with regard to other neoplastic diseases except for the ones that have been cured for more than 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Pathological response rate | Assessed at the time of surgery of liver metastases (between weeks 17-20 from enrollment)
  Primary:
  - To evaluate the activity of the regimen with regards to major/complete pathological response. Major/complete pathological response is measured by pathologist in terms of tumor regression grade (TRG) as described by Rubbia-Brandt L, Annals of Oncology 2007 (percentage of vial residual cells 0-10%).

SECONDARY OUTCOMES:
RECIST Response rate | Available at week 9 after enrollment
  - Response rate according to RECIST vers. 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Filippo de Braud, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Mi, Italy